CLINICAL TRIAL: NCT00845182
Title: Effect of Pioglitazone With and Without Exenatide on Body Weight, Fat Topography, Beta Cell Function, and Glycemic Control in Type 2 Diabetic Patients
Brief Title: Effect of Pioglitazone and Exenatide on Body Weight and Beta Cell Function
Acronym: PIO-EX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC2007243H
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes; Healthy; Impaired Glucose Tolerance
Keywords: Type 2 diabetes pathogenesis, thiazolidinediones; impaired glucose tolerance; Incretins; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Pioglitazone; Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pioglitazone (Active Comparator): Pioglitazone: 15 Patients will be randomized to Pioglitazone only arm
  Interventions: Drug: Pioglitazone
- Exenatide (Experimental): Exenatide: 15 subjects will be randomized to receive Exenatide
  Interventions: Drug: Exenatide
- Drug Pioglitazone and Drug Exentatide (Experimental): Pioglitazone and Exenatide: 15 subjects will be randomized to Pioglitazone and Exenatide
  Interventions: Drug: Pioglitazone and Exenatide

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg/day for 1 month and then 45 mg/day for 5 months
  Other Names: ACTOS
  Arms: Pioglitazone
Drug: Exenatide — Exenatide 5mcg twice daily for 1 month, then 10mcg twice daily for 5 months
  Other Names: BYETTA
  Arms: Exenatide
Drug: Pioglitazone and Exenatide — Pioglitazone 30mg daily for 1 month and then 45mg daily for 5 months and Exenatide 5mcg twice daily for one month then 10mcg twice daily for 5 months
  Other Names: ACTOS; BYETTA
  Arms: Drug Pioglitazone and Drug Exentatide

SUMMARY:
Pioglitazone, a drug used in treatment of type 2 diabetes has been shown to improve insulin sensitivity in skeletal muscle, liver, and fat cells. Despite the beneficial effects of pioglitazone to improve insulin sensitivity and reduce cardiovascular disease in high risk type 2 diabetic patients, weight gain has been a limiting factor. Exenatide, another agent used for treatment of T2DM, improves glycemic control and promotes moderate weight loss. In this proposal we will examine the effect of combination therapy with pioglitazone plus exenatide on body weight, fat topography, beta cell function, glycemic control, and plasma lipid levels in subjects with type 2 diabetes mellitus compared to treatment with each drug separately. Assessment of beta cell function will be performed by measuring the maximal insulin secretory capacity using a maximal hyperglycemic stimulus combined with an intravenous arginine stimulus.

DETAILED DESCRIPTION:
The thiazolidinedione (TZD) class of drugs has been shown to improve insulin sensitivity in skeletal muscle, liver, and adipocytes and to have anti-inflammatory and cardioprotective effects. The beta cell function, measured by the insulin secretion/insulin resistance index during the OGTT, improves significantly. In the present study, we will perform a more definitive assessment of beta cell function in TZD-treated diabetic patients by measuring the maximal insulin secretory capacity using a maximal hyperglycemic stimulus combined with an intravenous arginine stimulus.

Despite the beneficial effects of pioglitazone to improve insulin sensitivity and reduce cardiovascular events in high risk type 2 diabetic patients, weight gain has been a limiting factor for primary care physicians even though pioglitazone treatment leads to a redistribution of fat out of muscle/liver/visceral area to subcutaneous fat.

Exenatide (Byetta) is 39 amino acid peptide which exhibits biological actions similar to GLP-1. In clinical trials exenatide reduces HbA1c by 1-1.2% in subjects with type 2 diabetes and promotes moderate weight loss which is sustained for up to 2 years.

In this proposal we will examine the effect of combination therapy with pioglitazone plus exenatide on body weight, fat topography, beta cell function, glycemic control, and plasma lipid levels in subjects with type 2 diabetes mellitus compared to monotherapy with each agent separately. We postulate that combination therapy will result in significant weight loss (in contrast to the weight gain which accompanies pioglitazone treatment) and have an additive, or even synergistic, effect to improve beta cell function and glycemic control in type 2 diabetic patients who are inadequately controlled on oral agent therapy with metformin alone, a sulfonylurea alone, or combination of metformin plus a sulfonylurea. We will also compare the insulin secretion in healthy control subjects (NGT, n=15) and subjects with impaired glucose tolerance (IGT, n=15) to evaluate the relative decline in beta cell function in T2DM compared to NGT and IGT subjects. NGT and IGT subjects will participate only in a OGTT and a Hyperglycemic clamp- they will not receive any medication.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients must be on diet therapy alone or diet plus a sulfonylurea, or diet plus metformin, or diet plus sulfonylurea/metformin and have a HbA1c ≥ 7.0%.
2. Patients must have the following laboratory values:

   Hematocrit ≥ 34 vol% Serum creatinine ≤ 1.8 mg/dl AST (SGOT) ≤ 2 times upper limit of normal ALT (SGPT) ≤ 2 times upper limit of normal Alkaline phosphatase ≤ 2 times upper limit of normal
3. Patients must have been on a stable dose of allowed chronic medications for 30 days prior to entering the study.
4. Body weight must be stable (± 3-4 pounds) over the three months prior to study
5. The normal healthy control group will be age, weight (BMI), and gender matched with the diabetic group and must have a normal OGTT according to ADA criteria.
6. Subjects with IFG/IGT will have a FPG (100-125mg/dl) and/or 2-h plasma glucose (140-199mg/dl) according to ADA criteria.

Exclusion Criteria:

1. Patients must not have type 1 diabetes.
2. Patients must not have a fasting plasma glucose of greater than 270 mg/dl or HbA1c > 10.0%.
3. Patients must not have received a thiazolidinedione or insulin for more than one week during the year prior to randomization.
4. Patients with a history of clinically significant heart disease (New York Heart Classification greater than class 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devjit Tripathy, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Barter Research Center, ALM VA Hospital, San Antonio, Texas, United States

REFERENCES:
- [Derived] Guardado-Mendoza R, Chavez AO, Jimenez-Ceja LM, Hansis-Diarte A, DeFronzo RA, Folli F, Tripathy D. Islet amyloid polypeptide response to maximal hyperglycemia and arginine is altered in impaired glucose tolerance and type 2 diabetes mellitus. Acta Diabetol. 2017 Jan;54(1):53-61. doi: 10.1007/s00592-016-0904-7. Epub 2016 Sep 13. PMID 27624579

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone and Exentatide: Pioglitazone and Exenatide: 15 subjects will be randomized to Pioglitazone and Exenatide
Period: Overall Study
Arm/Group | Pioglitazone | Exenatide | Pioglitazone and Exentatide
Started | 13 | 15 | 15
Completed | 10 | 11 | 9
Not Completed | 3 | 4 | 6
Not completed — Lost to Follow-up | 3 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Exenatide | Pioglitazone and Exentatide | Total
Number analyzed (Participants) | 13 | 15 | 15 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 15 | 42
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (5.7) | 54.3 (8.5) | 53.8 (9.8) | 54.2 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 9 | 11 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pioglitazone, Exenatide and Combined Pioglitazone and Exenatide on Body Weight
Description: Effect of Pioglitazone, Exenatide and combined Pioglitazone and Exenatide on body weight and beta cell function
Time Frame: baseline and 6 months
Population: we analyzed the weight at the end of study completion
Measure: Mean (Standard Deviation); unit: kg
Groups:
- PIOGLITAZONE: PIO therapy led to a weigh gain of 5.5 kg
- EXENATIDE: PIO therapy led to a weigh loss of 2.4 kg
- PIOGLITAZONE and EXNATIDE: Combinatiton of PIoglitazone and Exenatide led to weight gain of 2.7 kg
Arm/Group | PIOGLITAZONE | EXENATIDE | PIOGLITAZONE and EXNATIDE
Number analyzed (Participants) | 10 | 11 | 9
kg | 5.5 (7.3) | 2.4 (2.8) | 2.7 (4.4)
Statistical Analysis 1: Comparison: PIOGLITAZONE vs EXENATIDE vs PIOGLITAZONE and EXNATIDE; Test type: Superiority or Other; p < 0.05, ANCOVA
Statistical Analysis 2: Comparison: PIOGLITAZONE vs EXENATIDE vs PIOGLITAZONE and EXNATIDE; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: HbA1c
Description: change in HbA1c was measured before and after treatment in three groups
Time Frame: baseline and 6 months
Population: There was a greater improvement in HbA1c from baseline after combined treatment with Pioglitazone and Exenatide when compared with either therapy alone.
Measure: Mean (Standard Deviation); unit: percent point decrease from baseline
Arm/Group | Pioglitazone | Exenatide | Drug Pioglitazone and Drug Exentatide
Number analyzed (Participants) | 10 | 11 | 9
percent point decrease from baseline | 1.37 (0.68) | 1.09 (0.68) | 1.91 (1.20)

3. Secondary Outcome: Effect Pioglitazone, Exenatide, and Pioglitazone Plus Exenatide • Insulin Sensitivity • Inflammatory Cytokines • Glucagon and Free Fatty Acids • Plasma Lipids
Description: Effect pioglitazone, exenatide, and pioglitazone plus exenatide on
  * Insulin sensitivity
  * Inflammatory cytokines
  * glucagon and free fatty acids
  * plasma lipids measured over a 6 month period
Time Frame: 6 months
Population: Data were not collected for this analysis
Groups:
- Effect Pioglitazone, Exenatide, and Pioglitazone Plus Exenatid: Effect pioglitazone, exenatide, and pioglitazone plus exenatide on
  * Insulin sensitivity
  * Inflammatory cytokines
  * glucagon and free fatty acids
  * plasma lipids measured over a 6 month period
Arm/Group | Effect Pioglitazone, Exenatide, and Pioglitazone Plus Exenatid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for 6 months.
Arm/Group | Pioglitazone | Exenatide | Pioglitazone and Exentatide
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/12 | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=12) | Exenatide (N=15) | Pioglitazone and Exentatide (N=15)
weight gain (General disorders) | 2 (2) | 0 (0) | 1 (1) — 2 patients in the Pioglitazone had weight gain >10kg
nausea (General disorders) | 0 (0) | 1 (1) | 0 (0) — one patientin exenatide group had persistent nausea and dropped out

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No